CLINICAL TRIAL: NCT06981091
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Parallel-group Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of XH-S004 Tablets in Patients With Non-cystic Fibrosis Bronchiectasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-S004-201
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: Bronchiectasis; Active neutrophil elastase; Fibrosis
MeSH Terms: conditions — Bronchiectasis; Fibrosis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Participant Group (Experimental): Participants received XH-S004 20 mg once daily (QD) , for 24 weeks.
  Interventions: Other: XH-S004 20 mg
- Arm 2: Participant Group (Experimental): Participants received XH-S004 40 mg once daily (QD) , for 24 weeks.
  Interventions: Other: XH-S004 40 mg
- Arm 3: Participant Group (Placebo Comparator): Participants received the matching placebo once daily (QD) , for 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: XH-S004 20 mg — Administered once per day for 24 weeks.
  Arms: Arm 1: Participant Group
Other: XH-S004 40 mg — Administered once per day for 24 weeks.
  Arms: Arm 2: Participant Group
Other: Placebo — Administered once per day for 24 weeks.
  Arms: Arm 3: Participant Group

SUMMARY:
The purpose of this study is to find out if XH-S004 can reduce pulmanary exacerbation over a 24-week treatment duration in participants with non-cystic fibrosis bronchiectasis.

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, placebo-controlled, parallel-group study conducted in china, aimed at evaluating the efficacy, safety and tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of XH-S004 administered once daily for 24 weeks in participants with non-cystic fibrosis bronchiectasis (NCFBE).

This study plans to enroll 231 patients with bronchiectasis. Patients who sign the informed consent form will be screened according to the enrollment criteria, and randomly divided into 3 groups. Participants in groups 1 and 2 will receive different doses of XH-S004. Participants in group 3 will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the procedures and methods of this trial and sign a written informed consent form;
2. Male or female paticipants aged 18-85 years (inclusive) ;
3. Chest HRCT shows bronchiectasis affecting one or more lobes, and the condition is clinically diagnosed as non-cystic fibrosis bronchiectasis (clinical manifestations include chronic cough, significant productive cough, and/or intermittent hemoptysis, with or without varying degrees of polypnoea and other symptoms);
4. Based on medical history and the determination of the investigator , participants have at least 2 documented pulmonary exacerbations in the past 12 months before Screening;
5. Are current sputum producers with a history of chronic expectoration and able to provide a spontaneous sputum sample at screening visit (as described by the patient) ;
6. The body mass index (BMI) is ≥18 kg/m2 at screening;
7. Participants must ensure and agree that from 28 days prior to signing the informed consent form to 28 days after the final administration, women of childbearing potential, male participants, and their partners will use effective contraception methods other than oral drugs (e.g., condoms or intra-uterine contraceptive devices) and will not donate sperm or eggs during this period

Exclusion Criteria:

1. Have a primary diagnosis of chronic obstructive pulmonary disease (COPD) or asthma
2. Have bronchiectasis due to cystic fibrosis (CF), hypogammaglobulinemia, common variable immunodeficiency, or alpha1-antitrypsin deficiency
3. Are currently being treated for a nontuberculous mycobacterial lung infection, allergic bronchopulmonary aspergillosis, or tuberculosis
4. Have any acute infections, (including respiratory infections)
5. Patients who have previously received therapy with DPP1 inhibitors of the same class

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Time to the First Pulmonary Exacerbation Over 24-Week Treatment Period | Baseline (Day 1) to Week 24
  Time to first pulmonary exacerbation was calculated as the number of days from the date of randomization to the date of first documentation of an exacerbation. Pulmonary exacerbation was defined as having 3 or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics (EMBARC guideline) : 1. Increased cough 2. Increased sputum volume 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis.

SECONDARY OUTCOMES:
Incidence of pulmonary exacerbation as defined by EMBARC over 24-week treatment period. | Baseline (Day 1) to Week 24
  Time to first pulmonary exacerbation was calculated as the number of days from the date of randomization to the date of first documentation of an exacerbation. Pulmonary exacerbation was defined as having 3 or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics (EMBARC guideline) : 1. Increased cough 2. Increased sputum volume 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis.
Incidence of Pulmonary exacerbation as defined by investigators over 24-week treatment period. | Baseline (Day 1) to Week 24
  The definition of pulmonary exacerbation determined by investigator was defined as: Compared with previous symptoms, patient's current symptoms have worsened but not meet the EMBARC guideline-defined criteria for pulmonary exacerbation . However, the invetigator will have determined that oral/IV antibiotic therapy is required.
Change from baseline in forced expiratory volume in 1 second (FEV1) in pulmonary function test at week 24 after first drug administration. | At baseline and at week 24
  FEV1 was used to assess lung function and is the maximum amount of air that can be forced out in one second after taking a deep breath.
Change from baseline in Quality of Life Questionnaire - Bronchiectasis (QOLB) respiratory symptoms domain score at week 24 after first drug administration; | At baseline and at week 24
  The QOL-B is a validated, self-administered patient reported outcome (PRO) that assesses symptoms, functioning, and health-related (HR) QOL for participants with non-cystic fibrosis
Change From Baseline in Concentration of Active Neutrophil Elastase (NE) in Sputum | Baseline (Day 1) to Week 24
  The concentration of active NE in sputum, was measured by the difference between the pre-treatment concentration, on-treatment concentration and post-treatment concentration. In bronchiectasis, activation of neutrophils in the airway leads to release of NE which leads to damaged airway walls, mucus hypersecretion, exacerbated inflammation, which in turn affects neutrophil and macrophage functions, increasing the risk of infection. Negative change from Baseline indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital Affiliated to fudan univercity, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No